CLINICAL TRIAL: NCT04531345
Title: The Cytokine Status of Covid-19 Patients
Brief Title: Cytokine Status of Covid-19 Patients
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, Assoc. Prof., Istanbul Training and Research Hospital
Other Study IDs: Covid Cytokine
Record Dates: First submitted 2020-08-27; First posted 2020-08-28 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Covid19
Keywords: interleukin; cytokine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group: Patients with Covid 19 PCR (+) results
  Interventions: Diagnostic Test: Flow cytometric analysis
- Control Group: Healthy volunteers
  Interventions: Diagnostic Test: Flow cytometric analysis

INTERVENTIONS:
Diagnostic Test: Flow cytometric analysis — IL-1β, IFN-α2, IFN-γ, TNF-α, MCP-1 (CCL2), IL-6, IL-8 (CXCL8), IL-10, IL-12p70, IL-17A, IL-18, IL-23, IL-33 cytokine analysis of COvid-19 patients and healthy volunteers

SUMMARY:
COVID-19, spreading rapidly all over the world, causes serious morbidity and mortality. In severe COVID-19 infections, after pulmonary inflammation, cardiovascular organ failure, cytokine storm, hemophagocytosis, septic shock, develops due to uncontrolled hypoxia, and isolated organ failure turns into multi-organ failure. It is noteworthy that it causes lymphopenia in patients. In the studies, the blood levels of certain inflammatory cytokines, interleukin-1β,interleukin-6 and TNF-α, were evaluated. In addition, blood values of a limited number of cytokines were investigated similarly in a limited number of studies published in our country.

DETAILED DESCRIPTION:
The causative agent of coronavirus 2019 (COVID-19) disease, which started in Wuhan province of China in December 2019, was severe acute respiratory failure syndrome coronavirus 2 (SARS-CoV-2), which quickly spread all over the world and caused a pandemic. COVID-19 can cause death with symptoms such as fever, cough, muscle pain, shortness of breath, and pneumonia (1). Pulmonary pathology of COVID-19 is diffuse alveolar damage, focal reactive hyperplasia of pneumocytes with patchy inflammatory cells, intravascular thrombosis, monocyte, macrophage and lymphocyte infiltration into pulmonary spaces. Severe infiltration of pulmonary tissue affects alveolar gas exchange. In addition, cardiovascular morbidity, tachyarrhythmia and thromboembolic events are observed in 1/5 of the hospitalized patients with troponin elevation, which is closely related to mortality. In severe COVID-19 infections, after pulmonary inflammation, cardiovascular organ failure, cytokine storm, hemophagocytosis, septic shock, develops due to uncontrolled hypoxia, and isolated organ failure turns into multi-organ failure. It is noteworthy that it causes lymphopenia in patients. In the studies , the blood levels of certain inflammatory cytokines, interleukin-1β,interleukin-6 and TNF-α, were evaluated. In addition, blood values of a limited number of cytokines were investigated in a similar way in a limited number of studies published in our country.

We aimed to study IL-1β, IFN-α2, IFN-γ, TNF-α, MCP-1 (CCL2), IL-6, IL-8 (CXCL8), IL-10, IL-12p70, IL-17A, IL-18, IL-23, IL-33 at Covid 19 and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Covid 19 PCR (+) results

Exclusion Criteria:

* Cancer Patients
* Patients with known immunodeficiency
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who admitted to the emergency department with the complaint of respiratory failure, lymphopenia in blood tests and Covid 19 (+) in the PCR tests are case group.
  Also healty volunteers who don't have complaint of respiratory failure, lymphopenia in blood tests and Covid 19 (-) in the PCR tests are control group.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Cytokine levels of patients | 1 month
  IL-1β, IFN-α2, IFN-γ, TNF-α, MCP-1 (CCL2), IL-6, IL-8 (CXCL8), IL-10, IL-12p70, IL-17A, IL-18, IL-23, IL-33 levels

CONTACTS AND LOCATIONS:
Overall Officials: Ufuk Oguz Idiz, Assoc. Prof, Principal Investigator — Istanbul Training and Research Hospital
Locations (1):
- Istanbul Training and Reseach Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Channappanavar R, Perlman S. Pathogenic human coronavirus infections: causes and consequences of cytokine storm and immunopathology. Semin Immunopathol. 2017 Jul;39(5):529-539. doi: 10.1007/s00281-017-0629-x. Epub 2017 May 2. PMID 28466096
- [Background] Hu B, Huang S, Yin L. The cytokine storm and COVID-19. J Med Virol. 2021 Jan;93(1):250-256. doi: 10.1002/jmv.26232. Epub 2020 Sep 30. PMID 32592501
- [Background] Soy M, Keser G, Atagunduz P, Tabak F, Atagunduz I, Kayhan S. Cytokine storm in COVID-19: pathogenesis and overview of anti-inflammatory agents used in treatment. Clin Rheumatol. 2020 Jul;39(7):2085-2094. doi: 10.1007/s10067-020-05190-5. Epub 2020 May 30. PMID 32474885